CLINICAL TRIAL: NCT01946711
Title: A Pilot Study to Investigate the Efficacy and Safety of Buparid/PARI SINUS Versus Budes® Nasal Spray in the Therapy of Chronic Rhinosinusitis (CRS) With Polyposis Nasi in Adult Patients
Brief Title: Buparid/PARI SINUS Versus Budes® Nasal Spray in the Therapy of Chronic Rhinosinusitis With Polyposis Nasi
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12082.101
Record Dates: First submitted 2013-09-04; First posted 2013-09-20 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Rhinosinusitis; Chronic Polyposis
Keywords: CRS; polyposis
MeSH Terms: conditions — Rhinosinusitis | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buparid; Treatment A (Experimental): Buparid 1 mg budesonide/2 ml nebuliser solution
  Interventions: Drug: Budesonide
- Budes; Treatment B (Active Comparator): Budes® Nasal Spray 50 µg budesonide/pump
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Inhalation
  Arms: Buparid; Treatment A
Drug: Budesonide — Nasal spray
  Arms: Budes; Treatment B

SUMMARY:
The study should create data for the selection of a clinically relevant primary endpoint to assess the efficacy and safety of Buparid/PARI SINUS as compared to Budes Nasal Spray in the therapy of chronic rhinosinusitis (CRS) with polyposis nasi in adult patients. Ideally, the selected parameter should allow a correlation between an objective methodology and the clinical outcome of the study patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of chronic rhinosinusitis (CRS) with polyposis nasi grade I-III
* Patient with a PNIF of > 7 l/min separated for left and right side of the nose
* Patient's written informed consent
* Male or female,>= 18 years of age
* Patient is able to undergo nasal therapy without restrictions
* Capable of understanding the purpose and risk of the clinical trial
* Female patients with childbearing potential must have a negative urine pregnancy test prior to first IMP administration
* Patient has completed correctly the diary during the Wash-in Phase

Exclusion Criteria:

* Patients with cystic fibrosis
* Patients with polyposis nasi grade IV
* Patients with prior sinonasal surgery (exemption: polypectomy)
* Patients with primary ciliaritis
* Pregnant or breastfeeding women
* Patients with suspected active upper airway infection
* Receipt of an investigational drug as part of a clinical trial within 4 weeks prior to first administration of IMP
* Drug or alcohol abuse
* End-stage malignancies
* Known hypersensitivity to Budesonide
* Patients with oral steroid therapy within the last 4 weeks
* Patients with frequent epistaxis (> 2 per month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Becker, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (4):
- Germany (4):
  - University Göttingen, Göttingen
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
  - University LMU Munich, Munich
  - HNO-Zentrum Mangfall-Inn, Rosenheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 patients not randomised
Period: Overall Study
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buparid; Treatment A | Budes; Treatment B | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change of Inflammation of the Nasal Mucosa and Paranasal Sinus
Description: Inflammation of the nasal mucosa and paranasal sinus was assessed using the Lund-Mackay score based on magnetic resonance imaging. The score can take on values between 0 and 24 points, with higher values indicating more severe impairment. The outcome investigated is the intraindividual mean score of 2 independent raters assessing the same images.
Time Frame: Change from Baseline to Week 8
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 8 | 6
units on a scale | -2 [-3.5 to 2.5] | -0.8 [-3.5 to 1]

2. Secondary Outcome: Safety Assessment
Description: Treatment-emergent adverse events (AEs) Each participant has been monitored for adverse events up to 26 weeks. All patients withdrawn from the study will be followed-up for AEs or SAEs for further 2 weeks or 4 weeks, respectively.
Time Frame: up to 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 8 | 6
Participants | 5 | 4

3. Other Pre Specified Outcome: Health-specific Quality of Life
Description: Health-specific quality of life was assessed by means of the self-rated, 22-item Sino-Nasal Outcome Test (SNOT-22). The SNOT-22 total score has a (theoretical) range of 0 - 110 points, with higher scores indicating more severe impairment.
  Presented are the mean values of the SNOT-22 total score after 24 weeks minus value at day 0 (baseline).
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 8 | 6
score on a scale | 23.6 [19.7 to 27.6] | 14.4 [9.8 to 18.9]

4. Other Pre Specified Outcome: Nasal Obstruction
Description: Nasal obstruction was assessed using the method of rhinomanometry by measuring the positive nasal inspiratory flow (PNIF). For the assessment the subject had to inhale maximally through the nose three times and the highest value of flow rate was recorded after 4 weeks and 8 weeks of treatment.
Time Frame: 4 weeks / 8 weeks
Measure: Mean (95% Confidence Interval); unit: ml/sec
Arm/Group | Buparid; Treatment A | Budes; Treatment B
Number analyzed (Participants) | 8 | 6
ml/sec
  Mean flow rate after 4 weeks | 746 [462 to 1031] | 574 [267 to 881]
  Mean flow rate after 8 weeks | 755 [644 to 867] | 646 [527 to 765]

ADVERSE EVENTS:
Time Frame: Each participant has been monitored for adverse events up to 48 weeks. All patients withdrawn from the study will be followed-up for AEs or SAEs for further 2 weeks or 4 weeks, respectively.
Arm/Group | Buparid; Treatment A | Budes; Treatment B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buparid; Treatment A (N=8) | Budes; Treatment B (N=6)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Sensitive Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-02-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT01946711/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT01946711/SAP_001.pdf